CLINICAL TRIAL: NCT07218848
Title: ProSalud: A Health Promotion Project to Reduce Cancer Risk in Latinos Living in Rural/Agricultural Communities Within Moffitt's Catchment Area
Brief Title: ProSalud in Latinos Living in Rural/Agricultural Communities Within Moffitt's Catchment Area
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MCC-23665
Record Dates: First submitted 2025-10-16; First posted 2025-10-20 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ProSalud (Experimental): Aim 1: Quantitatively assess feasibility and acceptability of ProSalud and explore changes in cancer risk reduction behaviors.
  Aim 2: Qualitatively examine ways to optimize ProSalud. After Aim 1 follow-up is completed, we will recruit a subgroup of parent participants and conduct focus groups to further assess ProSalud with the goal of refining and optimizing our culturally tailored health promotion and cancer prevention workshop to best meet needs and preferences of Latino community members. Semi-structured focus group questions will derive from our quantitative findings in Aim 1.
  Interventions: Other: Aim 1 Workshops; Other: Aim 2 Focus Groups

INTERVENTIONS:
Other: Aim 1 Workshops — Eligible Latino parents of 6 to 12-years-old will participate in a one hour (hour and a half) workshop focused on increasing rural Latino community members' knowledge about modifiable behaviors, such as healthy eating, physical activity, and sun protection. Participants will complete a baseline assessment a week before the workshop and a 2-month follow-up assessment. The assessments will be administered by research staff in person or over Zoom/telephone and will assess the acceptability and feasibility of the workshop and key modifiable health behaviors associated with cancer risk reduction.
Other: Aim 2 Focus Groups — Parents for Aim 2 focus groups will be randomly selected from each of the Aim 1 cohorts from those completing all Aim 1 components. Participating parents in the focus groups will be asked semi-structured questions derived from Aim 1 quantitative findings. These questions will further assess the content presented in ProSalud to refine and optimize our culturally tailored health promotion and cancer prevention workshop to best meet the needs and preferences of Latino community members.

SUMMARY:
The purpose of the study is to find out if Latino families living in rural parts of Florida are interested in learning about cancer prevention through our ProSalud program and whether it helps them make healthier choices to lower their risk of cancer. The study will also gather people's opinions about the program to find ways to improve it in the future. For the first part of our study, Latino parents with children between the ages of 6 and 12 will be invited to take part in a one-hour (or one-and-a-half-hour) workshop. The workshop will teach about healthy habits like eating well, being active, and protecting skin from the sun. For the second part of the study, some parents who participated in the workshops will be randomly chosen to join a focus group. In the focus group, they'll be asked questions to help us make the workshop better and make sure it fits the culture, needs, and preferences of Latino families in rural communities.

ELIGIBILITY:
Inclusion and Exclusion Criteria:

* We will include adults of any age and sex who are parents of a 6- to 12-year-old child. Parents must speak Spanish and be able to read and write at the 4th-grade level.

Parents who speak English in addition to Spanish can also take part in the study, always considering that the workshop will be conducted in Spanish.

* Individuals who are wards of the state will be excluded from participation in this study.
* If a participant chooses not to take part at any point, they may do so without any consequences or loss of services provided through RCMA. This ensures that their rights are protected, and their decision will not affect their access to any services or support.
* We may, by chance, include students and employees. However, we do not plan on collecting information that would indicate any of these statuses. No wards will be included in the study. Wards will not be included as research participants. Because recruitment will happen through RCMA, we anticipate most participants to be socially and/or economically disadvantaged. Participation in this study is entirely voluntary.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-05-22 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Acceptability | 1 year
  Acceptability will be confirmed if ≥80% of enrolled participants indicate an intention to implement behavioral recommendations.
Demand feasibility and adherence | 1 year
  The study will be considered feasible if ≥75% of eligible parents approached to participate in the study agree to enroll.
Implementation feasibility | 1 year
  Implementation feasibility will be established if 100% of data collection is completed in the 1-year timeframe.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Kanetsky, MPH, PhD, Principal Investigator — Moffitt Cancer Center; Marilyn Stern, PhD, Principal Investigator — University of South Florida
Locations (2):
- United States (2):
  - Moffitt Cancer Center, Tampa, Florida
  - University of South Florida, Tampa, Florida